CLINICAL TRIAL: NCT04621552
Title: Comparison of Woven EndoBridge Device Sizing With Conventional Measurements and Virtual Simulation Using the Sim&Size Software: A Multi-Center Experience
Brief Title: Virtual Simulation for Woven EndoBridge Device Sizing
Acronym: VS-WEB
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0601
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Aneurysm; Intracranial Aneurysm
Keywords: Intracranial Aneurysm; WEB; virtual simuation; SARS-CoV-2; Unruptured and Ruptrued intracranial aneurysms
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: WEB embolization — Treatment of intracranial aneurysms with WEB with the use of the virtual simulation before implantation of the device

SUMMARY:
Selection of the appropriate size of the device is mandatory during aneurysm treatment with a WEB. The Investigators aimed to investigate if virtual simulation with Sim&Size software may have an impact on technical, angiographic, and clinical outcomes after WEB treatment. Data from two large-volume centers were collected and compared (January 2017-January 2020). Virtual simulation was systematically adopted in one center, while conventional sizing was used in the other one. Outcomes were the duration of intervention, the radiation dose (mGy), the number of corrective interventions for inappropriate WEB size, the number of WEBs not deployed, angiographic occlusion, and complications. Univariate and multivariate linear models were adopted.

DETAILED DESCRIPTION:
Flow disruption with Woven EndoBridge (WEB) is an innovative treatment that has been evaluated in several prospective and retrospective studies1-3. The efficacy and safety of this strategy has been largely proved, and nowadays, indications for WEBs are progressively enlarged. Appropriate sizing of the device is the key factor for treatment with a WEB. Undersized devices may lead to insufficient coverage of the aneurysm neck and inadequate filling of the volume of the sac, lowering the angiographic success. On the other hand, an excessively oversized WEB may cause an unwarranted protrusion into the parent vessel, increasing the risk of ischemic events. The conventional approach for WEB sizing is based on two-dimensional digital subtraction angiography (2D-DSA), adding 1mm to the average width (to assure good wall apposition), and subtracting 1mm to the average height of the aneurysm (to adjust for the longitudinal increase caused by the horizontal compression)4. However, the operator has to anticipate the behavior of the device, predicting tridimensional modifications of the WEB in relation to the volume and shape of the aneurysm dome and neck. Accordingly, appropriate WEB sizing could be difficult and may require experience. Data about software-based simulation to predict changes after device implantation have been reported for flow diversion and braided stents5-7. The Sim&Size software (Sim&Cure, Grabels, France) is able to perform virtual sizing before WEB deployment using pre or per-operative three-dimensional rotational angiography (3D-RA) acquisition. The virtual simulation helps to select the most appropriate size of the device, predicting the behavior of the WEB inside the aneurysm dome, and the surface of the WEB apposition, anticipating protrusion over the neck or inappropriate coverage of the ostium. This multicenter study aimed to explore if the use of the Sim&Size software during endovascular embolization of intracranial aneurysms with WEB devices was associated with measurables procedural advantages compared with conventional sizing methods.

The primary investigated outcomes were 1) the median duration of the intervention; 2) the median radiation dose; 3) the need of corrective interventions; and 4) the number of WEBs opened but finally not deployed because of the inappropriate size of the device.

The secondary investigated endpoints were 1) the overall rate of complications (peri-procedural and long-term adverse events); 2) the morbidity rate (complications associated with permanent change of the clinical and neurological status of the patient); and 3) short-term (6 months) and long-term (12 months or more) aneurysm occlusion and WEB-shape change ("compaction") (decrease in height of the device or a deepening of the proximal and distal concave recesses during follow-up9 based on non-subtracted images)

ELIGIBILITY:
Inclusion criteria:

- Patients > 18 years treated with WEB for intracranial aneuryms

Exclusion criteria:

* Patients <18 years
* no eligibility for treatment with WEB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years treated with WEB for an intracranial aneurysms
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Median duration of the intervention | 1day
  the median duration of the intervention
Median radiation dose | 1 day
  the median radiation dose
Need of corrective interventions | 1 day
  the need of corrective interventions
number of WEBs opened | 1 day
  the number of WEBs opened but finally not deployed because of the inappropriate size of the device.

SECONDARY OUTCOMES:
Overall rate of complications | 1 day
  the overall rate of complications (peri-procedural and long-term adverse events)
morbidity rate | 1 day
  the morbidity rate (complications associated with permanent change of the clinical and neurological status of the patient)
Rate of Aneurysm occlusion | 6 months and 12 months
  short-term (6 months) and long-term (12 months or more) aneurysm occlusion
WEB-shape change | 6 months and 12 months
  WEB-shape change ("compaction") (decrease in height of the device or a deepening of the proximal and distal concave recesses during follow-up9 based on non-subtracted images).

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cagnazzo, MD PhD, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Cagnazzo F, Marnat G, Ferreira I, Daube P, Derraz I, Dargazanli C, Lefevre PH, Gascou G, Riquelme C, Morganti R, Berge J, Gariel F, Barreau X, Costalat V. Comparison of Woven EndoBridge device sizing with conventional measurements and virtual simulation using the Sim&Size software: a multicenter experience. J Neurointerv Surg. 2021 Oct;13(10):924-929. doi: 10.1136/neurintsurg-2020-017060. Epub 2020 Dec 23. PMID 33361275